CLINICAL TRIAL: NCT06731257
Title: Virtual Ward-Assisted Very earLy dIschArge of Low-rIsk STEMI patieNTs: the VALIANT-STEMI Trial
Acronym: VALIANT-STEMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CD24/163181
Record Dates: First submitted 2024-12-06; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Cardiovascular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): For the standard group and study participants the clinical records will be reviewed to check if any primary or secondary endpoints were met. They will be contacted at 30 days for a telephone consultation after the index event (time from when patient was admitted), and they will be asked to fill in a patient satisfaction questionnaire
- study group (Other): Patients who are randomised to the study group will receive a blood pressure monitor and instructions on how to use the device and transfer data to the study team. The study nurses will contact the patient every day for 3 days following their discharge and perform an virtual ward round assessment by telephone (see table). This will determine whether the patient continues to be monitored via the virtual ward, or whether they need to be referred to the clinical team. They will be issued with an emergency contact number out of hours (coronary care unit LGI) and the nursing hub will operate from 8am to 5pm 7 days a week. They will be referred to the community cardiac rehabilitation service whilst on the pathway.
  Interventions: Other: virtual ward early discharge

INTERVENTIONS:
Other: virtual ward early discharge — Patients who are randomised to the study group will receive a blood pressure monitor and instructions on how to use the device and transfer data to the study team. The study nurses will contact the patient every day for 3 days following their discharge and perform an virtual ward round assessment by telephone (see table). This will determine whether the patient continues to be monitored via the virtual ward, or whether they need to be referred to the clinical team. They will be issued with an emergency contact number out of hours (coronary care unit LGI) and the nursing hub will operate from 8am to 5pm 7 days a week. They will be referred to the community cardiac rehabilitation service whilst on the pathway.
  Arms: study group

SUMMARY:
Observational studies have suggested that early discharge (24hrs with follow up virtually by telephone) of patients who are low risk and have had successful treatment following ST elevation myocardial infarction is safe. This has not been tested in a randomised controlled trial. In this trial the study team propose to identify low risk patients and randomise them to usual care or early discharge and follow up virtually by telephone. The primary endpoint would be readmission to hospital or all cause death up to 30 day following the event. If the outcome is positive, the study will assist early discharge of patients, reduce length of stay, potentially improve patient well being and have positive financial implications for the health service

ELIGIBILITY:
Inclusion Criteria:

* Successful revascularisation following STEMI
* Zwolle score <=3
* No bystander disease awaiting inpatient intervention at the time of screening or consent (so if they have had intervention to a bystander vessel before this they would be eligible)

Exclusion Criteria:

* Haemodynamic instability (Killip class >I)
* Left ventricular ejection fraction <45%<40%
* Sustained ventricular or atrial arrhythmias requiring intervention
* No support at home or social or physical circumstances preventing early discharge
* Unable to use home monitoring equipment
* Unwilling to consent or follow instructions
* Patients visiting from out of our catchment area
* Out-of hospital cardiac arrest
* Patients repatriated to their local hospital within 24 hours
* New or worsening renal failure (i.e. creatinine >=1.5x baseline)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
30-day all-cause mortality or any rehospitalisation | 24-48 hours
  (time starts at admission of patient). No randomised controlled trials (RCTs) have compared 24-48 hours discharge to >48 hours discharge in low-risk STEMI patients. To the knowledge there has been a prior meta-analysis included 5 RCTs comparing discharge at 48 to 72 hours versus >72 hours and this was found to be safe(4). The 30-day event rate of any hospitalisation or all-cause death that was available from 3 RCTs was 31/489 (6.3%) in the routine care arm and 21/515 (4.1%) in the early discharge arm. For a non-inferiority design, assuming an event rate of 6% in the routine care arm and 4% in the very early discharge arm and a non-inferiority margin of 2.5%, 290 patients would be needed in each arm to provide 80% power, at 5% significance level. To allow for approximate 3-4% drop-out rate, it is intended to recruit 600 patients in total

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospital NHS Trust, Leeds, United Kingdom